CLINICAL TRIAL: NCT05912140
Title: TRACE2: Development of a New Tool for the Evaluation of the Trunk Aesthetics in Patients with Scoliosis
Brief Title: Assessment of Trunk Aesthetics: Development of a New Tool
Acronym: TRACE2
Status: Active, not recruiting | Type: Observational
Sponsor: Istituto Scientifico Italiano Colonna Vertebrale (Other)
Responsible Party: Sponsor
Other Study IDs: TRACE2
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Adolescent Idiopathic Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Trunk Aesthetic Clinical Evaluation
  Interventions: Other: TRACE 2

INTERVENTIONS:
Other: TRACE 2 — The first version of TRACE2 will be retrospectively verified through its application by experts on 150 photos of scoliosis patients who agreed to use the material produced for clinical use for retrospective research. Both intra-operator and inter-operator repeatability will be evaluated and a first Rasch analysis will be performed.
  The new version of TRACE2 (TRACE2.2) obtained following the retrospective validation on the photos will be verified prospectively through its application by the experts on 150 patients in specialist medical examination. Both intra-operator and inter-operator repeatability will be evaluated and further Rasch analysis will follow. On the basis of the results obtained from the analysis, the new TRACE2 scale (TRACE2.3) will then be applied to a further 150 patients, its intra- and inter-operator repeatability will be calculated and a final Rasch analysis will be performed to arrive at the final version of the scale (TRACE2.4).

SUMMARY:
Scoliosis is a three-dimensional deformity of the spine and the trunk. TRACE (Trunk Aesthetic Clinical Evaluation) is an aesthetics assessment tool for patients with scoliosis. It has been validated with Rasch analysis is easily usable in daily clinical practice. Despite this tool being more sensitive in detecting changes in aesthetics during treatment compared to other existing ones, its reliability is still low, probably due to the small number of elements that make up the rating scale.

This study aims to develop a new version of the TRACE tool by adding new items. The development of TRACE2 in a Rasch environment will ensure greater sensitivity and specificity of the scale assessment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of scoliosis
* age between 10 and 17 years old
* scoliosis >10° Cobb
* humps > 5° ATR

Exclusion Criteria:

* History of spinal surgery
* positive neurological assessment

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Adolescent with a diagnosis of scoliosis
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
TRACE2 | through study completion, an average of 1 year
  New version of the TRACE tool for the assessment of trunk aesthetics in patients with scoliosis

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Negrini, MD, Phd, Principal Investigator — Istituto Scientifico Italiano Colonna Vertebrale
Locations (1):
- ISICO, Milan, Mi, Italy

IPD SHARING:
Plan to Share IPD: Yes
Anonymous data will be deposited on an online repository